CLINICAL TRIAL: NCT03850717
Title: Retrospective Study on Safety of Acupuncture Treatments for Chronic Low Back Pain in 65 Years and Older in an Acupuncture Clinic From 2013 to 2018.
Brief Title: Safety of Acupuncture Treatments for Chronic Low Back Pain in Older Adults
Status: Completed | Type: Observational
Sponsor: McLean Center for Complementary and Alternative Medicine, PLC (Other)
Responsible Party: Sponsor
Other Study IDs: ATCMA 201901
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Chronic Low Back Pain; Older Adults
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Traditional Chinese Acupuncture: Use traditional acupuncture, stronger, deeper, "harder-acupuncture"
  Interventions: Device: acupuncture
- Japanese Acupuncture: Use traditional shallow, lighter acupuncture, "softer-acupuncture"
  Interventions: Device: acupuncture

INTERVENTIONS:
Device: acupuncture — insert in filiform needles into skin and other soft tissue to treat the illness or disorders

SUMMARY:
Acupuncture, along with other complementary and integrative treatments, is commonly used as a complementary or integrative therapy when treating a multitude of pain complaints, including chronic low back pain(CLBP). It has been practiced as a non-pharmacological therapy in the United States over one hundred years. Integrative pain management pilot programs have demonstrated impressive reductions in medications use, emergency room visits, and annual costs of healthcare. In fact, CLBP is one of the most common conditions treated in an acupuncturist's daily schedule. Based on acupuncturists' practice, CLBP has accounted for about 12% of patient visits in recent years. Most CLBP patients who come to acupuncturists' clinic are older adults. Investigators will retrospectively check the safety of acupuncture, i.e.side effects or adverse effects of acupuncture during treatments of CLBP in older adults in past 5 years.

DETAILED DESCRIPTION:
Back pain, especially low back pain (LBP), is one of the most common conditions for Americans to visit their physicians and therapists. In a recent survey, chronic neck and/or back pain was found to affect 54% of American adults in 2017. Another survey found that 32.5% of those 65 years and older suffer from back pain. Chronic low-back pain (CLBP) is defined by National Institutes of Health (NIH) as pain at the low back that persists for 12 weeks (3 months) or longer, even after an initial injury or underlying cause of acute low-back pain has been treated. About 20% of people affected by acute low-back pain develop CLBP with persistent symptoms at 1 year.

The inclusion criteria of CLBP in older adults:

Age: 65-80 years old. CLBP is defined as a back pain problem that has persisted for at least 3 months or has resulted in pain on at least half the days in the past 6 months. A minimum pain intensity score of 4 out of 10 on a visual analog scale (0 = no pain, 10 = most severe pain); ability of the participant to fully understand the trial procedure and the risks involved, communicate with the examiner, and comply with the protocol; provision of written informed consent for participation.

The exclusion criteria of CLBP in older adults:

Age: younger than 65. Pain mainly at legs; a history of spinal surgery; hip osteoarthritis; progressive neurological deficit or severe psychiatric or psychological disorders; serious spinal disorders, such as metastatic cancer, vertebral fracture, spinal infection, and inflammatory spondylitis; other contraindications for treatment, such as clotting disorders, use of anticoagulants or chemotherapy medications, and seizure disorders; presence of a device that could be affected by electromagnetic fields, such as a pacemaker; use of medications that could affect the trial results, such as corticosteroids and anticonvulsants, within the last week; participation in other clinical trials; ineligibility judged by a researcher.

For acupuncture in CLBP in older adults, one of public concerns is the safety of acupuncture. A thorough systematic review by Chan, et al. published in 2017 concludes that while some adverse events are reported, "all the reviews have suggested that adverse events are rare and often minor." These findings are consistent with prior studies. Some severe adverse events such as brain stem piercing, spinal lesions, infectious disease transmission, organ puncture, needle breaking and migrating, and death have been documented in other countries, but may be associated with provider competence and training, and could be avoided with sufficient regulations determining appropriate clinicians. Most of such severe adverse events are not within the scope related to the treatment in CLBP. There is no any specific acupuncture safety observation in treating CLBP in seniors. The aim of current study is retrospectively check all information documented related to side effects or adverse effects of acupuncture during treatments of CLBP in older adults in past 5 years. The treatments of acupuncture for CLBP are:

1. Acupuncture points (acupoints) or locations Use local points, in or near pain area, plus distant points. The local acupoints include Shenshu (BL23), Qihaishu (BL24), Dachangshu (BL25), and Guanyuanshu (BL26). These four pairs of points are located beside the L2-L5 spinal nerve foramen, while the CLBP may be related to L3-L5 nerves, erector spinae and associated fascia. Also use Yaoyan (EX-B-7). If the pain point (also called "tender point," "Ashi point" or "trigger point") is not located exactly at a traditional point location, consider the use of the tender point, instead of traditional point locations. If there are pain points (Ashi or trigger points) at gluteal muscles or the sacroiliac joint, add local points there as well. In clinical practice, 8-10 needles are used for these acupoints. The distant acupoints include Zusanli (ST36), Weizhong (BL40), Yanglingquan (GB34), Fengshi (GB31), and Sanyinjiao (SP6). I use up to 3 pairs of distal acupoints.
2. Needle sizes and needling technique Use 1.5-2.0 cun (40-50 mm), 30 or 32 gauge (G; 0.30 or 0.25 mm in diameter) filiform acupuncture needles. Occasionally, use 3.0 cun (75 mm), G30 needles for the gluteal muscle area (Cloud & Dragon, LEKON or EXPERT Traditional Acu Needles, manufactured and distributed by C.A.I. Corporation, USA). Prefer to treat patients in the prone position, inserting needles vertically (or slightly obliquely to the spinal foramen) about 1-1.5 cun (40-50 mm) deep, depending on patient size.
3. Inducing Deqi or not Use light Deqi technique [11]. That is, after inserting the needles, patients will feel some pressure or soreness at the local soft tissue area; at the same time, the acupuncturist will feel a pulling or pressure sensation from the inserted needle. Generally, do not use electric acupuncture for older adults with CLBP, due to the fact that such patients may have deficiency conditions. But use an infrared lamp to treat the low-back area during the acupuncture session. The acupuncture treatment lasts 45 min. After that, use light- to moderate-force suction cupping at the low-back pain area for 3-5 min.
4. Treatment duration Ideal treatment frequency or duration is 16-24 sessions: twice a week for 8-10 weeks, then once a week for 4 weeks, if possible. Most senior patients only have Medicare insurance, and in some cases, supplemental insurance; Medicare and supplemental insurance generally do not cover acupuncture. In the real world, senior CLBP patients have to pay out-of-pocket (give them some discount). Senior patients with CLBP may only choose to pay for 8-10 sessions, which may limit acupuncture's effectiveness.

One characteristic of CLBP in senior patients is that it may be due to a deficiency condition ("kidney deficiency" or "qi-blood deficiency"), which makes CLBP in seniors more difficult to treat than in younger adults. For this reason, one strategy of mine is using tonifying or strengthening acupoints: BL23, ST36, SP6, etc. Another strategy is to encourage patients to get more acupuncture sessions, such as 16-20 sessions, or say, after extensive treatments, then to get some tuning up sessions. In current investigator's practice, add Shenting (GV24), Yintang or ear Shenmen to calm patients' spirit, and help get a quicker effect in treating the older adults'CLBP.

In the United States, there has been no large-scaled acupuncture clinical trial of CLBP in older adults, especially focused on the real-world practice, therefore, there was no any safety evaluation study of acupuncture during the treatments of CLBP in older adults. In current studies, the investigators will check the CLBP senior (>65 years old) patients' files in past 5 years and find the detail safety information, i.e.side effects or adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age: 65-80 years old.
* CLBP is defined as a back pain problem that has persisted for at least 3 months or has resulted in pain on at least half the days in the past 6 months.
* A minimum pain intensity score of 4 out of 10 on a visual analog scale (0 = no pain, 10 = most severe pain);
* ability of the participant to fully understand the trial procedure and the risks involved, communicate with the examiner, and comply with the protocol;
* provision of written informed consent for participation.

Exclusion Criteria:

* Age: younger than 65.
* Pain mainly at legs;
* a history of spinal surgery;
* hip osteoarthritis; progressive neurological deficit or severe psychiatric or psychological disorders;
* serious spinal disorders, such as metastatic cancer, vertebral fracture, spinal infection, and inflammatory spondylitis;
* other contraindications for treatment, such as clotting disorders, use of anticoagulants or chemotherapy medications, and seizure disorders;
* presence of a device that could be affected by electromagnetic fields, such as a pacemaker;
* use of medications that could affect the trial results, such as corticosteroids and anticonvulsants, within the last week;
* participation in other clinical trials;
* ineligibility judged by a researcher.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: * age: 65 years or older;
  * both genders;
  * white, black and other nationalities.
  * with chronic low back pain.
  * Had at least one acupuncture treatment in McLean Center for Complementary and Alternative Medicine, PLC during the period of Dec. 31, 2013 to Dec.30, 2018.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-12-31 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
The rate of participates with bleeding | 2013-2018
  bruise in 3 levels: diameter<5mm, 6-10mm, >11mm

SECONDARY OUTCOMES:
The rate of participates with pain | 2013-2018
  3 levels: slight(<score 3), moderate (score 4-6), severe (score >7)
The rate of participates with fainting | 2013-2018
  3 levels: light-headed, slight faint, fainted.
The rate of participates with organ injury | 2013-2018
  Any organ injury-lung, heart, brain, liver, kidney, etc.
The rate of participates caused Infection | 2013-2018
  any infection related to acupuncture

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Y Fan, MD, PhD, LAc, Principal Investigator — McLean Center for Complementary and Alternative Medicine, PLC
Locations (1):
- McLean Center for Complementary and Alternative Medicine,PLC, Vienna, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
protect patients' personal information

REFERENCES:
- [Result] Fan AY, Ouyang H, Qian X, Wei H, Wang DD, He D, Tian H, Gong C, Matecki A, Alemi SF. Discussions on real-world acupuncture treatments for chronic low-back pain in older adults. J Integr Med. 2019 Mar;17(2):71-76. doi: 10.1016/j.joim.2019.01.005. Epub 2019 Jan 26. PMID 30738771
- [Result] Chan MWC, Wu XY, Wu JCY, Wong SYS, Chung VCH. Safety of Acupuncture: Overview of Systematic Reviews. Sci Rep. 2017 Jun 13;7(1):3369. doi: 10.1038/s41598-017-03272-0. PMID 28611366